CLINICAL TRIAL: NCT07289204
Title: FinnDiane LifeOne Study - Impact of Ageing on People With Type 1 Diabetes
Acronym: LifeOne
Status: Enrolling by invitation | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Folkhälsan Research Center (Unknown)
Responsible Party: Principal Investigator, Lena M. Thorn, Associate professor, Head physician, Helsinki University Hospital, Helsinki University Central Hospital
Other Study IDs: HUS/4387/2023
Record Dates: First submitted 2025-12-03; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Type 1; Healthy Ageing
Keywords: Aging; Healthy Aging; Diabetes Mellitus, Type 1; Prospective Studies; Cohort Studies; Geriatric Assessment; Finland
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetes: Participants of the Finnish Diabetic Nephropathy Study, age above 65 years.
- Controls: Age above 65 years, no diabetes with insulin therapy

SUMMARY:
Healthy aging refers to functional ability that enables well-being in older individuals. The focus thus shifts from chronological age to functional capacity and the individual's own experience of well-being. Type 1 diabetes is a chronic condition characterized by elevated blood glucose levels, which increases the risk of cardiovascular diseases and premature death. However, the life expectancy of individuals with type 1 diabetes has significantly improved due to advances in diabetes care.

There is limited research on aging with type 1 diabetes, and this study is at the forefront of addressing this gap by examining aging-and especially healthy aging-in type 1 diabetes from multiple perspectives. The goals are to investigate how individuals with type 1 diabetes age and what their functional capacity is compared to individuals without insulin-treated diabetes. The other aim is to identify factors in midlife that predict healthy aging in people with type 1 diabetes.

DETAILED DESCRIPTION:
Ageing with type 1 diabetes is an emerging challenge due to improved life-expectancy of people with type 1 diabetes. While those who survive to an older age are considered survivors, the many years with type 1 diabetes and the chronic dysglycaemia inevitably also has negative health impacts on people living with this chronic disease. With scarce research in this area, ageing in type 1 diabetes has been identified as a research gap.

With this study, the aim is to assess the impact of ageing in people with type 1 diabetes via thorough characterization of older adults with type 1 diabetes, in comparison to matched controls. This will be accomplished through a comprehensive assessment of the participants' metabolic profile, body composition, vascular health, autonomic function, and a geriatric assessment focusing on the functional ability of the participants. In addition, this study will assess what type of challenges older adults with type 1 diabetes face regarding self-management, diabetes care, and daily life.

This study is a sub-study of the national Finnish Diabetic Nephropathy Study, initiated in 1997 and including adults with type 1 diabetes. Individuals over 65 living in the Helsinki capital area will now be invited for a regular FinnDiane study visit, as well as an additional visit for a geriatric assessment. The aim is to study 300 FinnDiane study participants and recruit a minimum of 100 matched controls. This cohort will be prospectively followed with a revisit after three to five years.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the Finnish Diabetic Nephropathy Study
* Type 1 diabetes
* With age above 65 years
* Informed consent provided

Exclusion Criteria:

* Age below 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants of the Finnish Diabetic Nephropathy (FinnDiane) Study living in the Helsinki capital area. Controls will be recruited from spouses to match for sex and socioeconomic factors.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Healthy ageing in people with type 1 diabetes mellitus | From initial enrollment in the FinnDiane Study until the LifeOne follow-up visit after three to five years.
  Key Characteristics and Clinical Implications of healthy aging in individuals with type 1 diabetes mellitus

SECONDARY OUTCOMES:
Physical capacity | From initial enrollment in the FinnDiane Study until the LifeOne follow-up visit after three to five years.
  The locomotor domain of the individual's intrinsic capacity, based on the framework for healthy ageing.
Cognitive function | From initial enrollment in the FinnDiane Study until the LifeOne follow-up visit after three to five years.
  The cognitive domain of the individual's intrinsic capacity, based on the framework for healthy ageing.
Psychological well-being | From initial enrollment in the FinnDiane Study until the LifeOne follow-up visit after three to five years.
  The psychological domain of the individual's intrinsic capacity, based on the framework for healthy ageing.
Vitality | From initial enrollment in the FinnDiane Study until the LifeOne follow-up visit after three to five years.
  The vitality domain of the individual's intrinsic capacity, based on the framework for healthy ageing.
Sensory function | From initial enrollment in the FinnDiane Study until the LifeOne follow-up visit after three to five years.
  The sensory domain of the individual's intrinsic capacity, based on the framework for healthy ageing.

CONTACTS AND LOCATIONS:
Locations (1):
- HUS Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Individual-level data for the study participants are not publicly available because of the restrictions due to the study consent provided by the participant at the time of data collection. Researchers may propose collaboration to research the individual level data with correspondence with the lead investigator.